CLINICAL TRIAL: NCT00224510
Title: A Mulitcentre, Double-blind, Randomised, Fixed-dose Evaluation of the Safety and Efficacy of Lamictal (Lamotrigine) Compared to Placebo as an add-on Therapy to Lithium or Another Mood Stabiliser in the Treatment of Bipolar Depression, Followed by Long-term Prevention of Relapse and Recurrence of Depression and/or Mania in Patients With Bipolar Disorder
Brief Title: A Study To Investigate The Antidepressant Effect Of Lamotrigine In Patients With Bipolar Disorder Using Lithium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCA30905
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Bipolar Disorder; Bipolar Depression
Keywords: bipolar disorder bipolar depression lamotrigine
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lamotrigine

SUMMARY:
This is a study that, in the first 16 weeks, investigates whether lamotrigine versus placebo offers effect on depressive episodes for patients with bipolar disorder (also known as manic depressive disorder) who use lithium. In the following 50 weeks it is investigated whether these patients experience effect on their depressive and/ or (hypo)manic episodes.

DETAILED DESCRIPTION:
A Multicentre, Double-Blind, Randomised, Fixed-Dose Evaluation of the Safety and Efficacy of Lamotrigine (Lamictal®) compared to placebo as add-on therapy to lithium in the Treatment of Bipolar Depression followed by Long-term Prevention of Relapse and Recurrence of Depression and/or Mania in Subjects With Bipolar Disorder

ELIGIBILITY:
Inclusion criteria:

* Patients with bipolar disorder (type I or type II) currently suffering from depression that is at least moderate in severity according to a psychiatrist.
* Currently using lithium.
* Female subjects can't be pregnant or become pregnant during the study.

Exclusion criteria:

* Actively suicidal.
* Rapid cyclers.
* Suffering from significant personality disorders.
* Alcohol or substance dependent or abusive.
* Suffering from significant physical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2002-08 (Actual); Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Score on the MADRS depression rating scale at week 8 compared to baseline

SECONDARY OUTCOMES:
Scores on various mood rating scales and safety measurements at week 16 and between week 16 and week 68 compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (28):
- Netherlands (24):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Amersfoort
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Bennebroek
  - GSK Investigational Site, Blaricum
  - GSK Investigational Site, Delft
  - GSK Investigational Site, Dordrecht
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Flushing
  - GSK Investigational Site, Gouda
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Leiden
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Raalte
  - GSK Investigational Site, Retranchement
  - GSK Investigational Site, Rosmalen
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Tilburg
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Weert
  - GSK Investigational Site, Zwolle
- Spain (4):
  - GSK Investigational Site, Alava
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Valencia

REFERENCES:
- [Background] Poster presented at the APA congress, US, 2007 (Lamotrigine as add-on to lithium in bipolar depression) and the 5th European Stanley Conference on Bipolar Disorder in Barcelona, 2006)
- [Background] van der Loos ML, Mulder PG, Hartong EG, Blom MB, Vergouwen AC, de Keyzer HJ, Notten PJ, Luteijn ML, Timmermans MA, Vieta E, Nolen WA; LamLit Study Group. Efficacy and safety of lamotrigine as add-on treatment to lithium in bipolar depression: a multicenter, double-blind, placebo-controlled trial. J Clin Psychiatry. 2009 Feb;70(2):223-31. doi: 10.4088/jcp.08m04152. Epub 2008 Dec 30. PMID 19200421
- [Derived] van der Loos ML, Mulder P, Hartong EG, Blom MB, Vergouwen AC, van Noorden MS, Timmermans MA, Vieta E, Nolen WA; LamLit Study Group. Efficacy and safety of two treatment algorithms in bipolar depression consisting of a combination of lithium, lamotrigine or placebo and paroxetine. Acta Psychiatr Scand. 2010 Sep;122(3):246-54. doi: 10.1111/j.1600-0447.2009.01537.x. Epub 2010 Feb 5. PMID 20136801